CLINICAL TRIAL: NCT04046601
Title: Diagnosis of Early Barrett's Neoplasia and Esophageal Squamous Cell Neoplasia by Electrical Impedance Spectroscopy in Human Tissue
Brief Title: Impedance Spectroscopy in Esophageal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sana Klinikum Offenbach (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Barrett08/2019
Record Dates: First submitted 2019-08-04; First posted 2019-08-06 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Cancer of Esophagus
Keywords: impedance, Barrett´s cancer, early detection of cancer
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Intervention Model Description: Observation group: patient who are planned for endoscopic resection because of known esophageal cancer. Immediately after retrieval the resected specimens will be investigated for their electrical impedance properties. The results of the impedance measurement are compared to the histological results.
Masking Description: no masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Impedance (Experimental): every resected tissue will measured by an impedance probe
  Interventions: Device: impedance

INTERVENTIONS:
Device: impedance — After endoscopic resection of early esophageal cancer, the tissue will be measured by an impedance probe between 10Hz-1000000Hz, 20mV. 8 gold electrodes have been integrated to the probe. The impedance will be measured in different ways between the elctrodes. There will be 10 measurements in total for each specimen.

SUMMARY:
Detection of early esophageal cancer in surrounding normal tissue can be challenging even for experienced examiners. The early detection is essential to determine the following treatment. Early stages of esophageal cancers can be treated by endoscopic resection whereas advanced neoplasia might lead to an Operation of the esophagus. Diagnosis is made usually by biopsies of suspicious lesions or untargeted quadrant biopsies. The electrical properties in inflammatory tissue and cancer can be sensed by electrical bioimpedance technique.

The aim of this study is to compare the impedance probe with the histological result and to investigate the feasibility of the new technique in detection of esophageal cancer.

DETAILED DESCRIPTION:
Detection of early esophageal cancer in surrounding normal tissue can be challenging even for experienced examiners. The early detection is essential to determine the following treatment. Early stages of esophageal cancers can be treated by endoscopic resection (ER) whereas advanced neoplasia might lead to esophagectomy. Diagnosis is made usually by biopsies of suspicious lesions or untargeted quadrant biopsies. The electrical properties in inflammatory tissue and dysplasia can be sensed by electrical bioimpedance technique. The aim of this study is to compare the impedance probe with the histological result and to investigate the feasibility of the new technique in detection of esophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

Known esophageal cancer and planned for endoscopic resection

Exclusion Criteria:

1. Missing consent / agreement
2. Patient in bad condition for endoscopy or endoscopic resection
3. Patients with coagulopathy or anticoagulative medication which is a contraindication for endoscopy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2019-10-09 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-15 (Actual)

PRIMARY OUTCOMES:
impedance | 10 min
  value of 17 different frequencies in ohm

SECONDARY OUTCOMES:
differences in impedance | 10 min
  Differences in electrical impedance properties between different stages of early esophageal cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Mate Knabe, MD, Principal Investigator — Sana Klinikum Offenbach
Locations (1):
- Sana Clinic Offenbach, Offenbach, Hesse, Germany

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: SAP, Analytic Code
Time Frame: 6 month
Access Criteria: Data access request will be discussed by an internal board . Requestors will be required to sign a Data Access Agreement.

REFERENCES:
- [Derived] Blosser S, May A, Welsch L, Ast M, Braun S, Velten T, Biehl M, Tschammer J, Roeb E, Knabe M. Virtual Biopsy by Electrical Impedance Spectroscopy in Barrett's Carcinoma. J Gastrointest Cancer. 2022 Dec;53(4):948-957. doi: 10.1007/s12029-021-00703-0. Epub 2021 Sep 24. PMID 34559362